CLINICAL TRIAL: NCT03810014
Title: Malaria Diagnostic Testing and Conditional Subsidies to Target ACTs in the Retail Sector: the TESTsmART Trial AIM 1
Acronym: TESTsmART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Moi University (Other); Clinton Health Access Initiative, Nigeria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00100425; 1R01AI141444-01 (NIH)
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Malaria; Febrile Illness
Keywords: rapid diagnostic test (RDT); Artemisinin combination therapy (ACT); Conditional subsidy; Private retail sector
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: A factorial design will be used to test two ACT subsidy levels and two RDT subsidy levels. The unit of randomization will be the individual customer. Using scratch cards, participants will be randomized, in a 1:1:1:1 ratio, to one of four study arms:
  1) No subsidy for RDT (price to consumer=$0.40); 100% ACT subsidy (price to consumer=$0) // 2) No subsidy for RDT (price to consumer=$0.40); 67% ACT subsidy (price to consumer= $0.10-0.40, dependent upon patient age) // 3) 50% subsidy for RDT (price to consumer=$0.20); 100% ACT subsidy (price to consumer=0) // 4) 50% subsidy for RDT (price to consumer=$0.20); 67% ACT subsidy (price to consumer=$0.10-0.40, dependent upon patient age)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): The subsidy levels for participants randomly assigned to Arm 1 are: No subsidy for RDT (price to consumer=$0.40); 100% ACT subsidy (price to consumer=0).
  Interventions: Other: Conditional ACT subsidy, Arm 1 levels
- Arm 2 (Experimental): The subsidy levels for participants randomly assigned to Arm 2 are: No subsidy for RDT (price to consumer=$0.40); 67% ACT subsidy (price to consumer=$0.10-0.40, dependent upon patient age).
  Interventions: Other: Conditional ACT subsidy, Arm 2 levels
- Arm 3 (Experimental): The subsidy levels for participants randomly assigned to Arm 3 are: 50% subsidy for RDT (price to consumer=$0.20); 100% ACT subsidy (price to consumer=0).
  Interventions: Other: Conditional ACT subsidy, Arm 3 levels
- Arm 4 (Experimental): The subsidy levels for participants randomly assigned to Arm 4 are: 50% subsidy for RDT (price to consumer=$0.20); 67% ACT subsidy (price to consumer=$0.10-0.40, dependent upon patient age)
  Interventions: Other: Conditional ACT subsidy, Arm 4 levels

INTERVENTIONS:
Other: Conditional ACT subsidy, Arm 1 levels — The subsidy levels for participants randomly assigned to Arm 1 are: No subsidy for RDT (price to consumer=$0.40); 100% ACT subsidy (price to consumer=0).
  Arms: Arm 1
Other: Conditional ACT subsidy, Arm 2 levels — The subsidy levels for participants randomly assigned to Arm 2 are: No subsidy for RDT (price to consumer=$0.40); 67% ACT subsidy (price to consumer=$0.10-0.40, dependent upon patient age).
  Arms: Arm 2
Other: Conditional ACT subsidy, Arm 3 levels — The subsidy levels for participants randomly assigned to Arm 3 are: 50% subsidy for RDT (price to consumer=$0.20); 100% ACT subsidy (price to consumer=0).
  Arms: Arm 3
Other: Conditional ACT subsidy, Arm 4 levels — The subsidy levels for participants randomly assigned to Arm 4 are: 50% subsidy for RDT (price to consumer=$0.20); 67% ACT subsidy (price to consumer=$0.10-0.40, dependent upon patient age)
  Arms: Arm 4

SUMMARY:
The TESTsmART Trial consists of two main aims. The overall goal of the two aims is to investigate the impact of malaria rapid diagnostic test (mRDT) subsidies and conditional artemisinin combination therapy (ACT) subsidies on the testing and treatment behavior of participants seeking care for their febrile illness in the private retail sector. Conditional ACT subsidies are discounts on quality-assured ACTs which are linked to the results of a malaria rapid diagnostic test administered at the retail outlet; only participants with a positive test will have access to an additional discount on a quality-assured ACT.

The main objective of Aim 1 of this study is to identify a combination of conditional ACT and RDT subsidies that maximizes the proportion of participants that choose to have a malaria diagnostic test before taking a drug. The investigators will test two levels of conditional ACT subsidy (100% subsidy versus ~67% subsidy) and two levels of RDT subsidy (0% subsidy and 50% subsidy) in a factorial designed experiment. Because dose size and therefore the price of an ACT course are dependent upon patient age, the ACT subsidy amount will also be scaled with patient age. These subsidy levels were chosen to keep the estimated program cost of the combined subsidy within $0.30-0.60 USD per person (assuming 100% testing uptake and between 20-40% of participants having a positive RDT). These estimates represent an upper bound since testing is unlikely to reach 100%. Current subsidy levels for ACT costs the program between 1.30-2.50 USD per treatment, with more than a third of that investment spent on individuals without malaria.

Individuals presenting to a retail outlet for a treatment of a fever or suspected malaria illness will be randomized to one of the four groups in equal proportions. A total of 840 participants will be enrolled (210 per arm). Their choices concerning uptake of testing and drug purchase will be recorded. The main outcome will be the proportion of participants that choose to take a test. Secondary outcomes include the proportion of participants who adhered to the results of the RDT among those who were tested (used ACT when positive and did not use an ACT when negative or without a test). The results of this study will be used to inform the subsidy levels in the intervention for Aim 2 of this trial.

DETAILED DESCRIPTION:
RATIONALE:

From previous studies and implementation experiences, we know that consumption of ACTs increases as the price declines. Declining prices of ACTs create a trade-off between access and targeting; lower prices improve uptake of effective therapies by those with malaria but also increase inappropriate use by those without malaria. Curbing inappropriate use and targeting ACTs to malaria cases requires parasitological diagnosis which is virtually absent in the retail sector. It has also been shown that RDTs can be safely deployed in the retail sector. Most clients will agree to have an RDT if it is free. However, uptake of RDTs is sensitive to the price of the RDT. Previous work has not specifically evaluated the relationship between the price of the drug and the price of the test, but available evidence suggests that uptake of the RDT is sensitive to the price of the ACT as well.

In this work, we will link these two commodities through a diagnosis-dependent ACT subsidy. Access to the additional ACT subsidy depends on having a positive RDT. What we need to understand before scaling up a conditional subsidy is how the price of these two commodities should be related. Should the conditionally-subsidized ACT be less expensive than the RDT? Must the RDT be considerably less expensive than the retail price of ACT in order to motivate people to purchase a test?

OBJECTIVES:

In this study (Aim 1) we will use an individually-randomized experiment conducted among customers at medicine retail outlets to identify the combination of RDT subsidy-level and conditional ACT subsidy-level that maximizes uptake of diagnostic testing. We choose to focus on diagnostic testing because this is the first step to achieving the downstream goals of ACT targeting and rational use.

STUDY DESIGN:

We will use a factorial design to test two ACT subsidy levels and two RDT subsidy levels. The unit of randomization will be the individual customer.

STUDY POPULATION:

This study will be carried out in a sample of retail shops that carry quality-assured ACTs in our study area in western Kenya. Ten shops will be randomly selected to participate in the study. The study population will be any individual presenting to the shop with a malaria-like illness. Children older than 1 year of age are eligible to be enrolled provided they are physically present and accompanied by a parent or legal guardian. Customers with a prescription from a health facility, who have already received a malaria diagnostic test or who have already taken antimalarials prior to coming to the outlet will be excluded. Individuals who have signs of severe disease will be excluded and referred immediately to a health facility for care.

STUDY PROCEDURES:

A research assistant (RA) will be stationed at participating outlets on random days in order to avoid influencing treatment seeking behavior - in other words, to avoid attracting customers because of the study team's presence. The RA will obtain consent and offer participants a scratch card with a secret subsidy offer that will be revealed after the participant is enrolled. Using the scratch card, the participants will be randomized, in a 1:1:1:1 ratio, to one of four study arms: 1) No subsidy for RDT (price to consumer=$0.40); 100% ACT subsidy (price to consumer=0) // 2) No subsidy for RDT (price to consumer=$0.40); 67% ACT subsidy (price to consumer=$0.40) // 3) 50% subsidy for RDT (price to consumer=$0.20); 100% ACT subsidy (price to consumer=0) // 4) 50% subsidy for RDT (price to consumer=$0.20); 67% ACT subsidy (price to consumer=$0.10-$0.40, dependent on patient age).

These four arms represent a 2x2 factorial experiment.

If the participant chooses to purchase a test at their assigned price (subsidy level), the outlet will collect the money and the RA will perform the test. (RAs have been trained in RDTs and blood safety and have conducted thousands of RDTs. If the test is positive, the participant is entitled to an additional discount on their ACT purchase according to their group identified on the scratch card. If the test is negative, the participant may purchase any medicine they choose, including a regularly-priced ACT. Those who opt not to purchase an RDT may continue with their transaction as they choose, including purchasing a regularly-priced ACT.

The outlet attendant will sell the medicines to the customer, including a discounted ACT, if eligible. The study team will reimburse the outlet the difference between the retail price and the discounted price.

The RDTs selected for the study will be a World Health Organization (WHO) approved product that exceed 95% sensitivity and 95% specificity for Plasmodium falciparum [Malaria Rapid Diagnostic Test Performance, Round 1-5, WHO 2014].

STUDY OUTCOME MEASURES:

The primary outcome for Aim 1 is the customer's decision to purchase an RDT (yes/no). Using the 2x2 factorial design we will separately evaluate the effect of RDT price (2 levels) and of conditional ACT subsidies (2 levels) on the primary outcome.

The main secondary outcome is the proportion of tested participants who are adherent to the test result among those tested. Adherence is defined as taking a quality-assured ACT if the RDT is positive or taking another drug (or no drug) if the test is negative. We will also measure the proportion of people who purchase a full-price ACT among those who do not use an RDT.

SAMPLE SIZE:

We estimated the sample size required in each of the four study arms for a design with equal numbers of individuals allocated to each arm and where we wish to detect a 15-percentage point increase in RDT testing between an unsubsidized RDT compared to a subsidized RDT and to detect a 10 percentage-point difference in testing uptake between a partially and a fully subsidized ACT (conditional on a positive RDT) with at least 90% power and 5% chance of a two-tailed Type I error for each of the two comparisons. To do so, we estimate that we will need 210 subjects per arm (total=840).

ENROLLMENT AND FOLLOW UP:

All participants will be screened and enrolled on the day they visit the outlet. Data collection will be brief and will be completed on the same day. Participants will be screened as they arrive, enrolled if eligible and willing, tested if they choose and then allowed to proceed with their transaction at the outlet. Upon completion, they will be briefly interviewed again before leaving. Because the interaction with the participant is short and completed in one encounter, we expect minimal loss to follow-up (for example, participants leaving before the final questions).

ELIGIBILITY:
Inclusion Criteria:

* Participants with fever or history of fever or malaria like illness
* Individual with malaria-like illness must be present at recruitment
* 1 year of age or older

Exclusion Criteria:

* Any individual with signs of severe illness requiring immediate referral
* Individuals who have taken an antimalarial in the last seven days, including for the current illness
* Individuals who already have a prescription from a facility or medical provider
* Pregnant women will be enrolled and offered an mRDT, but will be advised to seek treatment through a health care provider.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 842 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy P O'Meara, PhD, Principal Investigator — Duke University
Locations (1):
- Moi University, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saran I, Laktabai J, Menya D, Woolsey A, Turner EL, Visser T, O'Meara WP. How do malaria testing and treatment subsidies affect drug shop client expenditures? A cross-sectional analysis in Western Kenya. BMJ Open. 2022 Dec 6;12(12):e066814. doi: 10.1136/bmjopen-2022-066814. PMID 36600353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was carried out in a random sample of twelve retail outlets in two sub-counties of rural western Kenya. Potential participants were approached by the research assistants as they sought services at the outlets. Participants were then offered a scratch card with masked arm assignment, which randomized them to one of four study arms in a 1:1:1:1 ratio, each arm with a different combination of two different RDT prices and two different conditional ACT prices using a 2x2 factorial design.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Started | 215 | 204 | 210 | 213
Completed | 213 | 202 | 210 | 211
Not Completed | 2 | 2 | 0 | 2
Not completed — Pregnancy | 2 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Six pregnant women were excluded from baseline characteristics and all following analysis because they didn't meet inclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Total
Number analyzed (Participants) | 213 | 202 | 210 | 211 | 836
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [11 to 45] | 28.5 [11 to 45] | 30 [16 to 43] | 31 [15 to 45] | 30 [13 to 45]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 97 | 96 | 92 | 103 | 388
  Male | 116 | 106 | 118 | 107 | 447
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 213 | 202 | 210 | 211 | 836
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 213 | 202 | 210 | 211 | 836
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Kenya | 213 | 202 | 210 | 211 | 836

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Purchase an mRDT (Malaria Rapid Diagnostic Test)
Description: This outcome will be evaluated once for each customer
Time Frame: At the end of a participant's visit to participating retail outlet, up to 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 213 | 202 | 210 | 211
Participants | 205 | 195 | 207 | 211
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4; (Arm 3 + Arm 4) vs (Arm 1 + Arm 2); Test type: Superiority; p = 0.01, Generalized estimating equations; Risk Difference (RD) = 2.50, 98% CI 2-sided [0.20 to 4.80]
Statistical Analysis 2: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4; (Arm 3 + Arm 4) vs (Arm 1 + Arm 2); Test type: Superiority; p = 0.012, Generalized estimating equations; Risk Ratio, log = 1.025, 98% CI 2-sided [1.002 to 1.049]
Statistical Analysis 3: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4; (Arm 1 + Arm 3) vs (Arm 2 + Arm 4); Test type: Superiority; p = 0.33, Generalized estimating equations; Risk Difference (RD) = -0.60, 98% CI 2-sided [-2.20 to 0.90]
Statistical Analysis 4: Comparison: Arm 1 vs Arm 2 vs Arm 3 vs Arm 4; (Arm 1 + Arm 3) vs (Arm 2 + Arm 4); Test type: Superiority; p = 0.332, Generalized estimating equations; Risk Ratio, log = 0.994, 98% CI 2-sided [0.979 to 1.009]

2. Secondary Outcome: Number of Participants With a Positive mRDT That Purchased an ACT (Artemisinin-based Combination Therapy)
Time Frame: At the end of a participant's visit to participating retail outlet, up to 1 hour
Population: Participants with a positive mRDT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 51 | 46 | 31 | 46
Participants | 47 | 39 | 24 | 40

3. Secondary Outcome: Number of Participants With a Negative mRDT That Did Not Purchase an ACT
Time Frame: At the end of a participant's visit to participating retail outlet, up to 1 hour
Population: Participants with a negative mRDT. 5 participants were not included due to missing ACT purchasing behavior; four in Arm 2 and one in Arm 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 154 | 145 | 175 | 165
Participants | 144 | 132 | 166 | 155

4. Secondary Outcome: Number of Participants That Did Not Purchase an mRDT and Did Not Purchase an ACT
Time Frame: At the end of a participant's visit to participating retail outlet, up to 1 hour
Population: Participants with no mRDT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Number analyzed (Participants) | 8 | 7 | 3 | 0
Participants | 4 | 5 | 3 | 0

ADVERSE EVENTS:
Time Frame: up to 1 hour
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
All-Cause Mortality (participants affected / at risk) | 0/213 | 0/202 | 0/210 | 0/211
Serious Adverse Events (participants affected / at risk) | 0/213 | 0/202 | 0/210 | 0/211
Other Adverse Events (participants affected / at risk) | 0/213 | 0/202 | 0/210 | 0/211

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT03810014/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT03810014/SAP_001.pdf